CLINICAL TRIAL: NCT07305532
Title: HARDWARE AND SOFTWARE DEVELOPMENT FOR PULMONARY MAGNETIC RESONANCE IMAGING USING INHALED INERT FLOURINATED GAS
Brief Title: ¹⁹F (Perfluoropropane) MRI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexei Ouriadov (Other)
Collaborators: St. Joseph's Health Care London (Other)
Responsible Party: Sponsor-Investigator, Alexei Ouriadov, PhD, professor, scientist, Western University
Organization: Western University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJHCF0001
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers - Male and Female
Keywords: 19F(perfluoropropane) MRI

STUDY DESIGN:
Intervention Model Description: Device: ¹⁹F (perfluoropropane) MRI
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ¹⁹F (perfluoropropane) MRI (Experimental): Participants will undergo pulmonary function tests, ¹⁹F (perfluoropropane) MRI at the visit.
  Interventions: Device: 19F(perfluoropropane) MRI

INTERVENTIONS:
Device: 19F(perfluoropropane) MRI — 19F(perfluoropropane) MRI is an emerging technique for imaging lung ventilation using inhaled, inert fluorinated gas. In contrast to proton-based MRI imaging, perfluoropropane gas is used as a contrast agent to directly visualize the airways, and thus ventilation. In this study, we aim to develop and evaluate an inert fluorinated gas-based MRI (19F MRI) technique to enhance non-invasive imaging in healthy adults without a history of acute or chronic respiratory disease.

SUMMARY:
"Healthy volunteers aged 18 to 85 will undergo ¹⁹F (perfluoropropane) MRI to support the development of imaging sequences, reconstruction algorithms, and hardware necessary for acquiring high-spatial resolution lung images. The study will also evaluate signal-to-noise ratio, contrast-to-noise ratio, spatial resolution, scan duration, and pulmonary gas exchange measurements derived from ¹⁹F (perfluoropropane) MRI.

DETAILED DESCRIPTION:
Briefly, during this two-hour visit, participants will provide written informed consent and then undergo:

1. Brief medical history and vital signs,
2. Full pulmonary function tests,
3. Proton MRI,
4. 19F(perfluoropropane) MRI, As part of the MRI, participants will inhale or 19F gas as a contrast agent to assess lung ventilation Spirometry will be performed at each visit according to American Thoracic Society (ATS) guidelines using MedGraphics Elite Series (MedGraphics Corporation. St. Paul, MN USA) and/or nDD EasyOne Spirometer (nDD Medical Technologies Inc. Andover, MA USA). Fractional exhaled nitric oxide (FeNO) will be measured using the NIOX VERO® (Circassia Pharmaceuticals Inc., Morrisville, NC, USA). All measurements will be performed at St Joseph's Healthcare London.

They will be placed in the 3T PET/MRI scanner with a coil fitted over their torso and chest. Hearing protection will be provided to muffle the noise produced by the 3D imaging gradient coils. A pulse oximeter lead will be used to monitor heart rate and oxygen saturation. MRI will be performed for up to a period of seven to ten minutes. All imaging will be performed in a "breath-hold" fashion. All participants will have supplemental oxygen provided via nasal cannula at a flow rate of at least two liters per minute during the scanning process. Logs and records of gas exposure will be maintained for every volunteer in this study.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must meet all of the following criteria:

1. Patient understands study procedures and is willing to participate in the study as indicated by the patient's signature.
2. Provision of written, informed consent prior to any study specific procedures.
3. Males and females aged 18 to 85 years.
4. Participant must be able to perform a breath-hold for 16s.
5. Participant has a BMI between 18 and 40
6. Participant must be able to perform reproducible pulmonary function tests (i.e., the 3 best acceptable spirograms have forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) values that do not vary more than 5% of the largest value or more than 100 ml, whichever is greater)
7. Participants are judged to be in stable health on the basis of medical history

Exclusion Criteria:

Participants fulfilling any of the following criteria are not eligible for inclusion in this study:

1. Patient has an MR incompatible implanted mechanically, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist).
2. In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI or CT, such as severe claustrophobia.
3. Participants who are pregnant, breastfeeding or have a positive pregnancy test at initial screening visit.
4. Participant is unable to perform spirometry maneuvers.
5. Participant is unable to perform MRI and CT breath-hold maneuvers.
6. Participant has a history of chronic or acute respiratory disease
7. FEV1 <70%
8. Participant has a history of cardiovascular disorders including coronary insufficiency, cardiac arrhythmias, severe hypertension (≥160 over ≥100)
9. Participant has a daytime room air oxygen saturation ≤ 92% ± 2% while supine

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Signal-to-noise ratio, Contrast-to-noise ratio, Image spatial resolution, and scan duration | 5 years
  The primary endpoints are to assess the necessary imaging sequences, reconstruction algorithms, and hardware to acquire high spatial resolution lung images from MRI,

SECONDARY OUTCOMES:
Ventilation Defect Percent (VDP) of the lung | 5 years
  VDP is a widely used noble gas MRI biomarkers that is calculated by normalizing ventilation defect volume to the thoracic cavity.
Fractional Ventilation (r) | 5 years
  Fractional Ventilation (r) is a quantitative imaging biomarker representing the fraction of gas volume in a lung region that is replaced by fresh inhaled air during a single breath. It is calculated using gas magnetic resonance imaging (MRI), where dynamic imaging tracks the wash-in and wash-out of inhaled gases (e.g., 19F (perfluoropropane)) within lung voxels. Fractional ventilation provides a regional measure of pulmonary ventilation efficiency and heterogeneity.

CONTACTS AND LOCATIONS:
Locations (1):
- St Joseph's Healthcare London, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified individual participant data supporting the results will be shared beginning 9 months after publication, available for up to 5 years. Access is open to researchers with approved proposals, subject to a data use agreement. Data will be shared via a secure platform upon approval